CLINICAL TRIAL: NCT06525454
Title: Feasibility and Acceptability of Individualized Automatic Target Coaching Message Based on the Metrics of Continuous Glucose Monitoring and Depressive Symptom
Brief Title: Individualized Automatic Target Coaching Message for Glycemic Management and Depressive Symptom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gyuri Kim, Samsung Medical Centor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-06-077
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Glucose

STUDY DESIGN:
Intervention Model Description: 1:2 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized coaching messages for glycemic management and depressive symptoms (Experimental)
  Interventions: Behavioral: Personalized coaching messages for blood glucose and emotions
- Treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: Personalized coaching messages for blood glucose and emotions — For six weeks, the intervention group will receive weekly personalized coaching messages for glycemic management based on blood data from continuous glucose monitors and bi-weekly personalized coaching messages for depression management based on depression questionnaires.
  Arms: Personalized coaching messages for glycemic management and depressive symptoms

SUMMARY:
This is a single-center, randomized, prospective, feasibility and acceptability trial in patients with type 1 diabetes. For six weeks, the intervention group will receive weekly personalized coaching messages for glycemic management based on blood data from continuous glucose monitors and bi-weekly personalized coaching messages for depression management based on depression questionnaires. The control group will remain on their current treatment and will not receive any intervention. The purpose of this trial is to evaluate the feasibility and acceptability of the clinical application of automated, personalized coaching messages for glycemic management and depressive symptom in people with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are determined to use continuous glucose monitoring based on their physician's medical judgment.
* Patients with type 1 diabetes, age 20-69 years old
* Currently receiving treatment with multiple insulin injection therapy
* Patients who have access to KakaoTalk via smartphone and are able to communicate with it
* Voluntarily agreed to participate in this clinical study.

Exclusion Criteria:

* Subjects using oral hypoglycemic agents
* Steroid and immunosuppressant users
* Subjects receiving anticancer medications
* Breastfeeding or pregnant patients
* Patients who do not voluntarily consent to the study
* Anyone deemed unsuitable by the investigator to participate in the study

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Time In Range | Week 6
  Derived from CGM

SECONDARY OUTCOMES:
Diabetes treatment satisfaction | Week 6
  DSTQ
Depressive symptoms | Week 6
  PHQ-9
Time In Tight Range | Week 6
  Derived from CGM
Time Above Range | Week 6
  Derived from CGM
Time Below Range | Week 6
  Derived from CGM
Coefficient of Variation | Week 6
  Derived from CGM
Glycemic Management Indicator | Week 6
  Derived from CGM

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No